CLINICAL TRIAL: NCT03570632
Title: Metformin for Preeclampsia Prevention in Pregnant Women With Type 1 Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maisa N. Feghali, MD (Other)
Responsible Party: Sponsor-Investigator, Maisa N. Feghali, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19060327
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1; Pregnancy in Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pregnancy in Diabetics | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention)
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Participants randomized to metformin will receive metformin in addition to standard treatment of diabetes during pregnancy
  Arms: Metformin

SUMMARY:
Although major advancements have been made in improving glycemic management in type 1 diabetes mellitus (DM), women entering pregnancy with type 1 DM continue to be at dramatically increased risk for adverse maternal and neonatal outcomes, including hypertensive disorders of pregnancy (HDP). At present, there is a lack of effective preventive interventions for HDP, which are associated with significant maternal and neonatal morbidity and mortality. Clinical and in vitro data have shown promise for metformin in prevention of HDP in non-diabetic women. Metformin has a reassuring fetal safety profile and has been well studied in type 1 DM outside of pregnancy. The hypothesis to be tested in this application is that compared to usual care, daily oral metformin therapy initiated prior to 20 weeks' gestation in women with type 1 DM reduces the frequency of HDP.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-50 years
* 12 0/7 and 19 6/7 weeks of gestation
* Diagnosed with type 1 DM prior to pregnancy.

Exclusion Criteria:

* Known allergy or adverse reaction to metformin
* Multiple gestation
* Abnormal obstetrical ultrasound suspicious for major congenital abnormality, known or suspected fetal aneuploidy
* Medical comorbidities that increase risk for metformin use: renal insufficiency (creatinine > 1.1 mg/dL), proteinuria (P:C >0.3 or 24-hour urine protein > 300 mg), active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes 3x above normal), inflammatory bowel disease (Crohn's and Ulcerative colitis), major hematologic disorder (including alloimmune and isoimmune thrombocytopenia).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant women are eligible to participate in the study
Enrollment: 60 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of hypertensive disorders of pregnancy | Delivery/End of pregnancy

SECONDARY OUTCOMES:
Home glucose levels throughout pregnancy | Weekly, throughout pregnancy from enrollment to delivery
Birthweight | Delivery/End of pregnancy
Neonatal morbidity | Delivery/End of pregnancy

OTHER OUTCOMES:
Gestational weight gain | At time of prenatal visits, throughout pregnancy from enrollment to delivery
Umbilical cord c-peptide | Delivery/End of pregnancy
Umbilical cord glucose | Delivery/End of pregnancy
Neonatal body composition | Delivery/End of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Maisa N Feghali, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No